CLINICAL TRIAL: NCT00207194
Title: Interactive Multirisk-Factor Intervention for HTN Blacks
Brief Title: Interactive Multirisk-Factor Intervention for Hypertension (HTN) Blacks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Principal Investigator, Julien Dedier, BUMC Faculty, Boston Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HL 69395
Record Dates: First submitted 2005-09-12; First posted 2005-09-21 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Automated Telephone Program (Active Comparator): The intervention was a totally automated, computer-based, interactive telephone counseling system called Telephone- Linked-Care, designed to monitor, educate, and counsel African-American adults with hypertension and to provide summary data regularly to the patient's primary care provider.
  Interventions: Behavioral: Automated Telephone Program; Behavioral: Health Behavior Education
- Health Behavior Education (Placebo Comparator): The comparator group received health education relating to the management of hypertension. Members of this group also received standard primary medical care.
  Interventions: Behavioral: Health Behavior Education

INTERVENTIONS:
Behavioral: Automated Telephone Program — The intervention incorporated principles of social cognitive theory, the transtheoretical model of behavioral change, and motivational interviewing, and was tailored to the user's values. Content was also adapted to cultural characteristics of culturally African-American adults (i.e., not Caribbean-American, Black-Hispanic, etc.). These participants also received the same health behavior education those in the control condition received.
  Arms: Automated Telephone Program
Behavioral: Health Behavior Education — Participants received a 75-page resource manual that described hypertension, listed dietary recommendations, heart healthy food recipes, and local resources for exercise, and provided information to support antihypertensive medication adherence. They received a 20-min education session based on the content of this manual, and were given a pedometer and a digital weight scale (Healthometer, model # HDR900KD01).

SUMMARY:
The aim of this study is to assess the efficacy of Telephone-Linked_Care for Hypertension Regimen Adherence in an African American population (TLC-HTN-AA). TLC-HTN-AA is a computer-based telecommunication system that will monitor, educate and counsel African American adults with hypertension on adherence to medication, diet, and exercise. The primary hypotheses are:

1. TLC-HTN-AA use will improve medication regiment adherence
2. TLC-HTN-AA will improve adherence to 3 healthy diet recommendations
3. TLC-HTN-AA will improve levels of regular exercise
4. Patients receiving TLC-HTN-AA will be more likely to become adherent to all 3 target regiments than patients in the control group

ELIGIBILITY:
Inclusion Criteria:

* a patient with a primary care provider at one of Boston Medical Center's Adult Primary Care Medical Practices or one of three HealthNet health centers participating in the study
* have a physician diagnosis of hypertension
* be African American by self-report
* be 35 years of age or older
* be prescribed at least one medication for hypertension
* have poorly controlled blood pressure
* be non-adherent to at least one hypertensive medication
* understand spoken English
* have a home telephone

Exclusion Criteria:

* patients for whom a medication, diet or exercise regiment adherence improvement or maintenance program would be inappropriate
* patients with a terminal illness
* patients with severe medical or psychiatric illness
* patients with cognitive difficulty

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 337 (Actual)
Dates: Start 2001-10; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
1-proportion of study subjects who achieve adequate adherence (greater than or equal to 80% of doses taken) at the end of the intervention period | 8 months
  Outcomes were assessed at baseline, 4 months, 8 months (the end of the study intervention) and 12 months.
2-consumption of more than 5 servings of fruits and vegetables a day, less than 30% of calories from fat, and less than 2400 mg of sodium a day at the end of the intervention period | 8 months
  Outcomes were assessed at baseline, 4 months, 8 months (the end of the study intervention) and 12 months.
3-adherence to CDC-ACSM recommendations for moderate intensity physical activity at the end of the intervention period | 8 months
  Outcomes were assessed at baseline, 4 months, 8 months (the end of the study intervention) and 12 months.

SECONDARY OUTCOMES:
1-TLC-HTN-AA use will reduce the mean blood pressure and the proportion of the treatment group having uncontrolled hypertension at the end of the intervention period | 8 months
  Outcomes were assessed at baseline, 4 months, 8 months (the end of the study intervention) and 12 months.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Friedman, MD, Principal Investigator — Boston Medical Center; Jeffrey Migneault, PhD, Study Director — Boston University
Locations (1):
- Medical Information Systems Unit/Boston Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Result] Migneault JP, Dedier JJ, Wright JA, Heeren T, Campbell MK, Morisky DE, Rudd P, Friedman RH. A culturally adapted telecommunication system to improve physical activity, diet quality, and medication adherence among hypertensive African-Americans: a randomized controlled trial. Ann Behav Med. 2012 Feb;43(1):62-73. doi: 10.1007/s12160-011-9319-4. PMID 22246660